CLINICAL TRIAL: NCT00820001
Title: Enhancing Long-Term Outcome in Child Behavior Disorders
Brief Title: Resources to Enhance the Adjustment of Children (REACH)
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, David Kolko, Professor of Psychiatry, Psychology, and Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH057727 (NIH)
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Cognitive Behavioral Therapy; Multimodal Treatment; Physiological Parameters; Hormone Concentration in pubertal development; Treatment as usual comparison
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acute Treatment Protocol Booster (Experimental): Child participants in this arm were initial participants enrolled in the parent study and randomized to receive the specialty treatment from study clinicians in either the clinic or community setting. In this continuation study, the participants were enrolled at the 36 month assessment and randomized to participate in the booster dose of treatment. The treatment provided in this arm includes specific booster treatment based on the 8 modules of the initial treatment study. Saliva samples were also collected 2 times in the lab and 2 times at home (once at bedtime, once at wake-up time) per initial voluntary saliva protocol at each timepoints to measure endocrine levels.
  Interventions: Behavioral: Booster Treatment
- Acute Treatment Protocol No-Booster (Experimental): Child participants in this arm were initial participants enrolled in the parent study and randomized to receive the specialty treatment from study clinicians in either the clinic or community setting. In this continuation study, the participants were enrolled at the 36 month assessment and randomized to participate in assessments only thus not receiving any additional booster treatment. Saliva samples were collected 2 times in the lab and 2 times at home (once at bedtime, once at wake-up time) per initial voluntary saliva protocol at each timepoints to measure endocrine levels.
  Interventions: Behavioral: No-Booster
- Treatment As Usual (Active Comparator): Child participants in this arm were initial participants enrolled in the parent study in the clinically referred Treatment As Usual comparison group. These participants were initially enrolled in treatment services with identified providers and received treatment services as provided in that community agency. In this continuation study, the participants were enrolled at the 36 month assessment and participated in the ongoing follow-up assessments only. Saliva samples were collected 2 times in the lab and 2 times at home (once at bedtime, once at wake-up time) per initial voluntary saliva protocol at each timepoints to measure endocrine levels.
  Interventions: Other: Treatment As Usual
- No Intervention Healthy Comparison (Other): The Healthy Control subjects enrolled initially in the parent study are incorporated in a related project designed to evaluate the role of biological measures in differentiating antisocial and normal children. All Healthy Control participants were initially matched to cases in the clinical sample (both the acute treatment and the clinically referred Treatment as Usual).
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Booster Treatment — Based on this collective evidence, booster treatment was designed to address three general goals: a) clarify key child and parent/family problems and family preferences regarding target problems, b) directly target and resolve these existing problems using the eight domains contained in the existing treatment protocol administered in the initial outcome study, and c) provide the family with clinical recommendations and information to promote the maintenance of skill developments in targeted domains or adaptive routines designed to prevent any further deterioration in clinical functioning. Thus, the clinician may provide a review of prior content or administer new material specifically for older adolescents, as needed, and will attempt to apply these skills to specific problematic situations identified by the family.
  Other Names: Modular Cognitive Behavior Therapy
  Arms: Acute Treatment Protocol Booster
Behavioral: No-Booster — All cases randomized to this condition will simply participate in all of the proposed routine assessments and will receive assessment feedback. Specifically, these families will be provided with a brief summary of the significant clinical findings obtained in their 36-month follow-up assessment (assessment feedback). Such an assessment was provided to clinicians in the original study in order to highlight specific areas in need of clinical attention based on a review of the normative data and clinical cutoffs available for each instrument. Selected information will be conveyed by phone to the participating parent/guardian in a straightforward manner followed by a discussion of some clinical recommendations designed to address these clinical problems. In addition, the parent/guardian will be provided with a listing of professionals who provide services appropriate for this age group and for children with similar problems.
  Other Names: No-Booster Comparison condition
  Arms: Acute Treatment Protocol No-Booster
Other: No intervention — No intervention was administered with this arm. Saliva samples were collected 2 times in the lab and 2 times at home (once at bedtime, once at wake-up time) per initial voluntary saliva protocol at each timepoints to measure endocrine levels.
  Other Names: Healthy Control Comparison Group
  Arms: No Intervention Healthy Comparison
Other: Treatment As Usual — All cases assigned to this arm simply participated in all of the proposed routine assessments.
  Other Names: Treatment As Usual clinical comparison.
  Arms: Treatment As Usual

SUMMARY:
This continuation study evaluates the long-term outcomes of multimodal, modular interventions with early-onset behavior disordered children and innovative methods to promote the maintenance and extension of treatment effects relating to ODD and CD. All participants originally enrolled in the "parent" clinical trial are being followed and those who initially received clinic or community based intervention from a study clinician were randomly assigned to either Booster or No-booster treatment condition. The treatment-as-usual (TAU) and Healthy Control participants were also followed through long-term follow-up assessments paralleling clinically referred participants. The study examines the short and long-term efficacy of booster treatment on clinical outcome, contextual variables, and service satisfaction/use.

DETAILED DESCRIPTION:
Child Conduct problems (CP), as found in Conduct Disorder (CD) and Oppositional Defiant Disorder (ODD), are common and chronic. Although laboratory research studies have yielded promising initial outcomes, follow-up effects are often not studied and, when they are evaluated, are often limited. Maintenance procedures have been generally administered after acute treatment in the form of periodic booster sessions to enhance long-term outcomes (Whisman, 1990). Although the conceptualization and application of maintenance therapies has been described frequently with adults, there is limited information regarding the role of maintenance treatment in child and adolescent psychotherapy (see Eyeberg, 1998). A few studies of booster treatments have reported the return of behavioral improvements (Baer, Williams, Osnes, & Stokes, 1984; McDonald & Budd, 1983; Patterson, 1974) and other improvements in conduct-disordered children (Lochman, 1992) and depressed adolescents (Clark et al., 1999), suggesting potential benefits in extending the durability of treatment effects. What is not yet known is the extent to which patients respond positively to a booster (maintenance) treatment condition that is administered after long-term (i.e., three-year) follow-up, one that is designed to reduce recurrence of behavioral dysfunction and the development of new forms of dysfunction during adolescence. The justification for this additional intervention derives from our initial findings and the young age of our sample, which, in most instances, has yet to traverse the period of heightened risk for delinquency.

Literature reviews highlight the importance of addressing at least three primary objectives in understanding the clinical response and long-term adjustment of children with ODD or CD. First, there is a need to document empirically the long-term effects of both specialty treatments and routine services during repeated follow-up assessments in an effort to document the maintenance of all initial treatment gains (Eyberg et al., 1998). Our preliminary findings suggesting the presence of both similarities and differences in the initial outcomes of our two specialty treatments (Community vs. Clinic protocols) supports the conduct of a long-term evaluation in order to determine whether these effects continue or change.

Second, our initial findings underscore the importance of determining the extent to which booster treatment sessions help to promote long-term maintenance or produce long-term preventive effects on some of the more common sequelae of ODD and CD. Booster treatment may be needed to deflect such children from unfolding trajectories toward increased antisocial behavior and multi-system impairments (Loeber et al., 1993). Thus, efforts to promote the long-term outcomes of follow-up in this population must be evaluated in an effort to understand the degree to which they show improvements in serious clinical dysfunction (recovery from Disruptive Behavior Disorders (DBD)) and/or show reductions in the development of new forms of dysfunction (deviant and delinquent activities) that may place these children at-risk for other adverse adolescent outcomes. The young age of this patient sample at the start of this competing continuation(8-16 yrs) may make it easier to demonstrate preventive effects.

Finally, the availability of only modest empirical evidence provides a compelling argument for evaluating potential predictors of each of the above-mentioned long-term follow-up outcomes based on a comprehensive battery of psychosocial (e.g., child, parent, and family adjustment) and biological (e.g., testosterone, cortisol) measures obtained upon study intake and treatment termination. Key predictors of treatment response include lower levels of child, parent, and family dysfunction, barriers to treatment, and SES (Kazdin, 1995; Kazdin & Wassell, 2000). We will also evaluate the role of contextual or other life changes in understanding treatment effects over the follow up period. Among the important contextual variables to be evaluated include changes in parental and family functioning, peer relationships, and school adjustment. Clearly, these variables may influence continued antisocial behavior at this young age. Thus, we will examine how contextual factors affect how well treatment effects hold as well as the real world impact of treatment on various life changes.

ELIGIBILITY:
All participants were enrolled in the initial "parent" study and criteria for initial enrollment included:

Inclusion Criteria:

1. males or females with an age of 6-11 years,
2. a DSM-IV diagnosis of CD or ODD,
3. residence with at least one parent/guardian;
4. intellectual level no less than two SD's below age norms; and
5. parent consent for participation.

Exclusion Criteria:

1. concurrent individual or family participation in a treatment program directed towards the child's disruptive disorders,
2. current psychosis, bipolar disorder, or MDD marked by significant vegetative signs,
3. suicidality with a plan or homicidality; or
4. substance abuse or an eating disorder.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2003-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Individualized child problem targets and externalizing behavior including functional impairment | Baseline for continuation (36 months into study participation) and at months 42, 48, 54, 66 (assessment timeline is inclusive of all assessments for parent and continuation trials)
Peer and Family Characteristics | Assessed at all follow-up timepoints including baseline (36 month assessment) and all subsequent follow-up assessments at months 42, 48, 54 and 66.
Parental Disfunction | Assessed at all timepoints including baseline (36 month) and follow-up assessments at months 42, 48, 54, and 66

SECONDARY OUTCOMES:
Teacher reports of child functioning | Assessed at all timepoints including baseline (36 month) and follow-up assessments at months 42, 48, 54, and 66
Child attentional and internalizing problems | Assessed at all timepoints including baseline (36 month) and follow-up assessments at months 42, 48, 54, and 66

CONTACTS AND LOCATIONS:
Overall Officials: David J Kolko, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bellefield Towers - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Kolko DJ, Dorn LD, Bukstein OG, Pardini D, Holden EA, Hart J. Community vs. clinic-based modular treatment of children with early-onset ODD or CD: a clinical trial with 3-year follow-up. J Abnorm Child Psychol. 2009 Jul;37(5):591-609. doi: 10.1007/s10802-009-9303-7. PMID 19221871
- [Result] Diler RS, Birmaher B, Axelson D, Goldstein B, Gill M, Strober M, Kolko DJ, Goldstein TR, Hunt J, Yang M, Ryan ND, Iyengar S, Dahl RE, Dorn LD, Keller MB. The Child Behavior Checklist (CBCL) and the CBCL-bipolar phenotype are not useful in diagnosing pediatric bipolar disorder. J Child Adolesc Psychopharmacol. 2009 Feb;19(1):23-30. doi: 10.1089/cap.2008.067. PMID 19232020
- [Result] Dorn LD, Kolko DJ, Shenk CE, Susman EJ, Bukstein O. Influence of treatment for disruptive behavior disorders on adrenal and gonadal hormones in youth. J Clin Child Adolesc Psychol. 2011;40(4):562-71. doi: 10.1080/15374416.2011.581614. PMID 21722028